CLINICAL TRIAL: NCT02122939
Title: An Open-label, Single Dosing Clinical Trial to Investigate the Pharmacokinetics and the Effect on ECG of Escitalopram After Oral Administration in Elderly Volunteers
Brief Title: A Clinical Trial to Investigate the Pharmacokinetics and the Effect on ECG of Escitalopram in Elderly Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, Associate professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ECTE
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — Escitalopram

ARMS (1):
- Escitalopram (Experimental)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram

SUMMARY:
An Open-label, single dosing clinical trial to investigate the pharmacokinetics and the effect on ECG of escitalopram after oral administration in elderly volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy subject aged 65 or older at screening
* A body weight in the range of 50 kg (inclusive) to 90 kg (inclusive) with BMI range of 19.0 to 28.0
* subjects who decide to participate voluntarily and write a informed consent form

Exclusion Criteria:

* subjects who have clinically significant disease of cardiovascular, respiratory, renal, endocrinological, hematological, gastrointestinal, neurological(central nervous system), psychiatric disorders or malignant tumor
* Subject judged not eligible for study participation by investigator

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Cmax, AUCinf, AUClast, Tmax, t1/2, CL/F | pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 32, 48 h post-dose

SECONDARY OUTCOMES:
QTc interval | pre-dose, 1, 4, 6, 8, 12, 24, 28, 32, 48 h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Chung, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital, Seongnam, Korea
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyounggi, South Korea